CLINICAL TRIAL: NCT05188560
Title: Efficacy of a Single Preoperative Administration of Action Observation Therapy Associated With Motor Imagery in Patients Undergoing Total Hip Arthroplasty.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 750
Record Dates: First submitted 2021-12-20; First posted 2022-01-12 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-01

CONDITIONS: Hip Osteoarthritis; Orthopedic Disorder
Keywords: Action observation therapy; motor imagery; Hip arthroplasty; functional recovery
MeSH Terms: conditions — Osteoarthritis, Hip; Musculoskeletal Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AOT+MI (Experimental): participants who, in addiction to standard rehabilitation program after surgery, underwent a single pre-operative training session of action observation therapy associated with motor imagery.
  Interventions: Other: Action observation therapy; Other: motor imagery
- Control group (No Intervention): Participants who was not subjected to any pre-operative activity. They received standard rehabilitation program after surgery too.

INTERVENTIONS:
Other: Action observation therapy — Subject is asked to observe videos with motor contents
  Arms: AOT+MI
Other: motor imagery — mental simulation of a motor task
  Arms: AOT+MI

SUMMARY:
Action Observation Therapy (AOT) and Motor Imagery (MI) are two rehabilitation approaches based on Mirror Neuron System (MNS). The MNS refers to a series of neurons able to activate both when one observes an action being performed or when one physically performs the action themselves. Previous studies reported that functional recovery is facilitated by asking patient observing videos with motor content (AOT) and after imagining (MI) the gestures observed. These rehabilitative apporach have been used in particular to promote functional recovery in patients with neuromotor problems, in particular in patients with stroke. To date, few studies have investigated the effectiveness of this therapeutic approach in functional recovery after orthopedic surgery and none of these applied AOT and MI in a single pre-operative session. The objective of the study is to verify whether a single administration consisting of two pre-operative sessions of AOT associated with MI can lead to an improvement of functional recovery in hip arthroplasty patients.

ELIGIBILITY:
Inclusion criteria:

* Total hip arthroplasty (THA) monolateral, first implant
* Locomotor autonomy with or without aids before surgery
* BMI (regular, overweight, Grade I obesity)
* No complications in surgery
* Orthopaedic prescription of tolerance load on the limb
* Autonomy with aids within the third post-operative day

Exclusion Criteria:

* Previous total hip replacement on contralateral hip
* Dementia or other conditions affecting patient's collaboration
* Unresolved clinical complications in the first two post-operative days
* Neurological, musculoskeletal or other disorders able to impact on functional recovery
* Visual or auditory deficits
* Total or partial revisions of THA
* Patients assigned to different groups hospitalized in the same room

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Changes in functional mobility using Timed Up and Go test (TUG). | Both groups will be evaluated the day before (T0) and 4 days after (T1) surgery.
  The primary outcome is to investigate whether a single administration consisting of two sessions of AOT and MI performed the day before the total hip arthroplasty may impact on functional recovery in the immediate post-operative period. Functional mobility will be evaluated with Timed Up and Go test.

SECONDARY OUTCOMES:
Changes in maximum gait speed | Both groups will be evaluated the day before (T0) and 4 days after (T1) surgery.
  Changes in maximum gait speed between and within groups will be evaluated with 10 meters-walking test (10 MWT).
Changes in pain using Visual Analogue Scale (VAS) | Both groups will be evaluated the day before (T0) and 4 days after (T1) surgery.
  Pain will be assessed with Visual Analogue Scale (VAS 0-10) ranging from 0 (absence of pain) to 10 (maximum pain)

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Clinico Humanitas, Rozzano, Milano, Italy